CLINICAL TRIAL: NCT05790642
Title: Vergleich Verschiedener Nicht-invasiver Verfahren Zur Pulswellenanalyse
Brief Title: Comparison of Different Non-invasive Methods to Assess Pulse Wave Analysis
Acronym: MULTI-PWA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: 202103Multi-PWA
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Blood Pressure; Arterial Stiffness; Arrythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Participants with sinus rhythm
  Interventions: Device: Pulse wave measurement and analysis
- Participants with atrial fibrillation
  Interventions: Device: Pulse wave measurement and analysis
- Participants with extra systoles
  Interventions: Device: Pulse wave measurement and analysis
- Participants with heart failure with reduced ejection fraction
  Interventions: Device: Pulse wave measurement and analysis
- Participants with mildly reduced or preserved ejection fraction
  Interventions: Device: Pulse wave measurement and analysis

INTERVENTIONS:
Device: Pulse wave measurement and analysis — Different contact-less and cuff-less pulse wave measurements will be used and compared to cuff-based reference method.

SUMMARY:
The primary goal of the study is to compare different methods for pulse wave measurement and analysis which are cuffless and contactless. The novel measurement tools will be compared to cuff-based reference methods.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* male or female sex
* signed informed consent.

Exclusion Criteria:

* acute sickness which influences hemodynamic parameters
* arm circumference is below or above the limits for the blood pressure of the reference method (i.e. below 20 or above 40 cm)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: general population
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2023-05-10 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure | 3 months
  Cuffless and contactless methods will be used to measure and analyze pulse wave velocity to estimate systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular examination center of the University Medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No